CLINICAL TRIAL: NCT05432518
Title: Biomarker and Tumor Cell Culture-Driven Pilot Trial for Treatment of Recurrent Glioblastoma
Brief Title: Pilot Trial for Treatment of Recurrent Glioblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBM-2022
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma; Recurrent Disease; Recurrent Glioblastoma
Keywords: Glioblastoma; Recurrent Disease; Recurrent Glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Afatinib; Dasatinib; palbociclib; Everolimus; olaparib

STUDY DESIGN:
Intervention Model Description: Open-label, pilot, umbrella trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients will receive one of the 5 study drugs based on their recurrent tumor mutation profile and their recurrent organoid response to these drugs:
  1. Afatinib
  2. Dasatinib
  3. Palbociclib
  4. Everolimus
  5. Olaparib
  Interventions: Drug: Afatinib; Drug: Dasatinib; Drug: Palbociclib; Drug: Everolimus; Drug: Olaparib

INTERVENTIONS:
Drug: Afatinib — Afatinib will be administered orally at a dose of 40 mg daily in patients with EGFR amplification.
  Other Names: Giotrif
Drug: Dasatinib — Dasatinib will be administered orally at a dose of 100 mg once daily in patients with PDGFR amplification.
  Other Names: Sprycel
Drug: Palbociclib — Palbociclib will be administered orally at a dose of 125 mg once daily in patients with CDK4 and CDK6 amplification.
  Other Names: Ibrance
Drug: Everolimus — Everolimus will be administered orally at a dose of 10 mg daily in patients with PI3K/PTEN/mTOR activated pathways.
  Other Names: Teva-everolimus
Drug: Olaparib — Olaparib will be administered orally at a dose of 300 mg twice daily in patients with TP53 mutation.
  Other Names: Lynparza

SUMMARY:
This will be a single-arm open-label prospective pilot feasibility trial recruiting 10 adult patients with recurrent glioblastoma who are assigned to receive the personalized study treatment based on the genetic profile of their recurrent GBM tumor resected at the time of surgery. It will be aimed to gather preliminary information on the study intervention and the feasibility of conducting a full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

1. Study participant has provided informed consent prior to initiation of any study specific activities/procedures.
2. Adult participants, male and female, aged ≥18 who have a pathologically confirmed IDH-wild type glioblastoma, with first or second progression of the tumor, after initial treatment with radiation therapy and temozolomide.
3. Recurrence is amenable to resection.
4. Performance status: ECOG ≤2.
5. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
6. Patients of childbearing potential must adhere to the contraception requirement from screening throughout the study period up to 180 days after the last dose of study intervention. Women/men of childbearing potential must have agreed to use two highly effective contraceptive methods. In addition to routine contraceptive methods such as condom use, oral contraceptive, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures.

   Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
7. Able to undergo brain MRIs.
8. Females must not be breastfeeding, throughout the study period up to 180 days after the last dose of study intervention.
9. Male patients should agree to not donate sperm during the study for at least 6 months until discontinuation of study drug.

Exclusion Criteria:

1. Patients with history of abnormal left ventricular ejection fraction (LVEF≤ 45%).
2. Pregnant, breast-feeding, unwilling/unable to comply with contraception requirements.
3. Patients unable to consent.
4. Abnormal (grade ≥2 CTCAE, version 5.0) laboratory values for hematology, renal, and liver function including:

   1. Hemoglobin <10,
   2. Neutrophils <1.5,
   3. Platelets <75,
   4. ALT/AST >3x ULN,
   5. Bilirubin >1.5 x ULN,
   6. eGFR <60
5. Patients with significant or recent gastrointestinal disorders with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption or severe diarrhea of any etiology) must be excluded from the clinical trial (Afatanib is not recommended in this patient population).
6. Patients with a history of ILD (interstitial lung disease) must be excluded.
7. Patients with severe hepatic impairment (Child Pugh C).
8. A significantly abnormal ECG (baseline QTcF interval > 450 msec).
9. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
10. Patients with known pre-existing pleural effusion.
11. Active hepatitis B or C infection and/or known history of HIV infection.
12. Has known psychiatric or substance abuse disorders that would interfere with compliance with the requirements of the trial.
13. Subject will not be available for protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge.
14. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks from the date of signing the informed consent form.
15. Patients who are hypersensitive to any ingredients in the formulation of the study drugs or their excipients.
16. Patients receiving active treatment for a different cancer.
17. If recent bacterial infection, patients need to have completed antibiotic course prior to commencing study drug.
18. If recent COVID-19 infection, patients must have recovered from it prior to commencing study drug.
19. Patients on strong CYP3A/p-gp inducers (for example, carbamazepine and phenytoin).

N.B. Only patients receiving SOC neurosurgery in Alberta, Canada are eligible to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of personalized GBM treatment based on molecular characterization of recurrent tumor | From date of initial consent to participate to the end of follow up period (24 months)
  Percentage of patients, interested in participating, consented and detected with target mutations and completed the treatment with one of the 5 study drugs

SECONDARY OUTCOMES:
Overall survival (OS) | From date of study drug administration until date of death from any cause (approximately 24 months)
  OS is calculated as the period from the day of starting administration of the study drug to the day of death from any cause.
Progression free survival (PFS) | From date of study drug administration until date of radiographic confirmed progression (approximately 2 years)
  PFS is calculated as the period from the day of starting administration of the study drug to the date that disease progression is confirmed by radiographic assessment and RANO criteria.
Quality of Life (QoL) EORTC QLQ-C30 | Baseline until the end of treatment
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Quality of Life (QoL) EORTC QLQ BN-20 | Baseline until the end of treatment
  Quality of Life measures are recorded according to EORTC QLQ BN-20 module, which is validated for brain tumor patients and measured as a unit of scale. This is a standard tool for assessing patient reported quality of Life along time during treatment. EORTC QLQ BN-20 (BN-20): 4 scales comprised of multiple items and 7 single items. All items are rated on a 4-point Likert-type scale, 1=not at all' to 4=very much, and linearly transformed to a 0-100 scale, higher scores indicating more severe symptoms.
  The scores across all time points were averaged to obtain the mean.

OTHER OUTCOMES:
Genomic and expression profiling | From date of initial consent to participate to end of follow up period (24 months)
  Number of patients for whom we were able to have genomic and expression profiling on their tissue samples and organoids
Organoid drug response | From date of initial consent to participate to end of follow up period (24 months)
  Number of patients for whom we can determine organoid drug response to study drugs
Correlation of genomic and expression profiling of tissue and organoid with the organoid's best drug response | From date of initial consent to participate to end of follow up period (24 months)
  Number of patients for whom the genomic and expression profiling of their tissue and organoid directly correlates to the organoid's best drug response

CONTACTS AND LOCATIONS:
Overall Officials: Paula de Robles, Principal Investigator — Arthur J.E. Child Comprehensive Cancer Centre
Locations (1):
- Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided